CLINICAL TRIAL: NCT01545310
Title: An Open-Label, Positron Emission Tomography (PET) Study to Evaluate the Brain 5 HT6 Receptor Occupancy by Single Doses of SLV354 in Healthy Male Subjects and Subjects With Stable Schizophrenia
Brief Title: A Positron Emission Tomography Study of SLV354 in Healthy Subjects and Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M12-700
Record Dates: First submitted 2011-12-15; First posted 2012-03-06 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (healthy), Group 2 (schizophrenia) (Experimental)
  Interventions: Drug: SLV354

INTERVENTIONS:
Drug: SLV354 — One dose of ABT-354
  Other Names: ABT-354

SUMMARY:
This open-label, Phase 1 study will investigate the 5-hydroxytryptamine 6 (5-HT6) receptor occupancy in the brain using positron emission tomography (PET) following single oral doses of SLV354. Up to 22 healthy male subjects and male subjects with stable schizophrenia, between 18-55 years of age are to complete the study.

DETAILED DESCRIPTION:
This is an exploratory, open-label PET study designed to examine the relationship between SLV354 plasma concentration and 5-HT6 receptor occupancy in the brain following single oral doses of SLV354 in healthy male subjects and male subjects with stable schizophrenia. A total of up to 22 subjects are to complete the study, including approximately 12 subjects with schizophrenia on a stable dose of an atypical antipsychotic medication. Within 60 days prior to the PET scan, subjects will be screened based on medical history, physical examination, vital signs, ECG, clinical laboratory tests, response to Columbia-Suicide-Severity Rating Scale (C-SSRS) and for schizophrenia subjects only, the diagnosis of schizophrenia based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR). Following Screening, eligible subjects will have a Magnetic Resonance Imaging (MRI) scan, unless one was performed within one year of the PET scan, to delineate the region of interest for the individual PET images. The radiotracer [11C]-QUICS will be used for the PET scans.

All subjects will receive a single oral dose of SLV354. Healthy subjects will have one PET scan prior to and two PET scans after administration of SLV354. Schizophrenia subjects will have two PET scans prior to and one PET scan after administration of SLV354.

ELIGIBILITY:
Inclusion Criteria

1. Male, age between 18 and 55 years, inclusive.
2. Body Mass Index 18 to 30 (healthy) and 18 to 38 (schizophrenia).
3. A condition of general good physical health.
4. Schizophrenia subjects must have a diagnosis of schizophrenia based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR).
5. Schizophrenia subjects must be on a stable dose of an atypical antipsychotic for at least 4 weeks prior to Screening.

Exclusion Criteria

1. Presence of a metal implant that would preclude a Magnetic Resonance Imaging (MRI) scan.
2. Radiation exposure for research purposes within the past year that will exclude participation in the study.
3. Significant current suicidal ideation within the past month as evidenced by Columbia-Suicide Severity Rating Scale (C-SSRS) completed at Screening.
4. History of psychiatric diseases or disorders (healthy subjects)
5. Unsuitable to receive SLV354 or the radiotracer, [11C]-QUICS.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Brain receptor occupancy | Study Day -1
  5-HT6 receptor occupancy and the relationship between SLV354 plasma concentrations and receptor occupancy
Brain receptor occupancy | Study Day 1
  5-HT6 receptor occupancy and the relationship between SLV354 plasma concentrations and receptor occupancy

SECONDARY OUTCOMES:
Pharmacokinetic profile | Up through Study Day 4
  Maximum observed plasma concentration (Cmax), time to Cmax (Tmax), area under the plasma concentration-time curve (AUC), terminal elimination half-life (t1/2), oral plasma clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Earle Bain, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 52162, New Haven, Connecticut, United States